CLINICAL TRIAL: NCT06373094
Title: A Single-center, Open-label, Single-dose Ascending Phase I Clinical Study Evaluating the Safety, Tolerability, and Pharmacokinetic Profile of HHT201 (Donepezil Dihydroxynaphthalate for Injection) in Healthy Subjects
Brief Title: A Single Dose Escalation Study of HHT201 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Synergy Pharmaceutical Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zhejiang Huahai Pharmaceutical Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DON102-CTP
Record Dates: First submitted 2024-03-19; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Single dose of 34 mg Donepezil Dihydroxynaphthalate for Injection.
  Interventions: Drug: Donepezil Dihydroxynaphthalate for Injection
- Group 2 (Experimental): Single dose of 68 mg Donepezil Dihydroxynaphthalate for Injection.
  Interventions: Drug: Donepezil Dihydroxynaphthalate for Injection
- Group 3 (Experimental): Single dose of 136 mg Donepezil Dihydroxynaphthalate for Injection.
  Interventions: Drug: Donepezil Dihydroxynaphthalate for Injection
- Group 4 (Experimental): Single dose of 204 mg Donepezil Dihydroxynaphthalate for Injection.
  Interventions: Drug: Donepezil Dihydroxynaphthalate for Injection
- Group 5 (Experimental): Single dose of 306 mg Donepezil Dihydroxynaphthalate for Injection.
  Interventions: Drug: Donepezil Dihydroxynaphthalate for Injection
- Group 6 (Experimental): Single dose of 408 mg Donepezil Dihydroxynaphthalate for Injection.
  Interventions: Drug: Donepezil Dihydroxynaphthalate for Injection

INTERVENTIONS:
Drug: Donepezil Dihydroxynaphthalate for Injection — HHT201 will be injected into the muscle of gluteus.
  Other Names: HHT201

SUMMARY:
The objective of this study is to evaluate the safety and pharmacokinetic profiles of HHT201 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy subjects, both male and female;
2. 20 years old ≤ 60 years old;
3. The weight of women is not less than 45 kg, the weight of men is not less than 50 kg, and the BMI is between 19 and 28 (including the upper and lower limits);
4. Understand and sign informed consent to participate in clinical trials voluntarily.

Exclusion Criteria:

1. Patients with a history of cardiovascular, respiratory, liver, kidney, endocrine system, digestive system, blood and lymphatic system, immune system, nervous system, skeletal system, psychiatric and other major diseases, who were judged not suitable for participation in this study;
2. Comprehensive physical examination, laboratory examination, vital signs, or past medical history are judged by clinicians to be abnormal and clinically significant;
3. ALT or Cr, BUN beyond the upper limit of normal values; Urine protein test results were "++";
4. Abnormal electrocardiogram (ECG) during the screening period had clinical significance, such as QTcF interval ≥450 ms in males and QTcF interval ≥470 ms in females, and the researchers considered it inappropriate to be included;
5. Those who had used CYP3A4 inhibitors such as ketoconazole, itraconazole, erythromycin, or CYP2D6 inhibitors such as fluoxetine and quinidine within 30 days before the screening period, or rifampicin, phenytoin sodium, and carbamazil equal liver drug enzyme inducers, or had taken any prescription drugs, over-the-counter drugs, Chinese herbs, vitamins, or other dietary supplements within two weeks before enrollment;
6. People who have taken food or drink (such as grapefruit) containing enzymes that can induce or inhibit liver metabolism within 1 week before the start of the trial;
7. People who have a history of severe allergy or have a history of allergy to two or more drugs, or to any of the components of Donepezil dihydroxynaphthoate for injection;
8. Patients with positive results of serum virology test [Hepatitis B surface antigen (HBsAg), Hepatitis Be antigen (HBeAg), hepatitis C virus antibody (HCV-IgG), human immunodeficiency virus (HIV) antibody, Treponema pallidum antibody (Anti-TP)];
9. Subjects with smoking history within 2 weeks prior to the screening period or positive results of urine cotinine test during the admission review period;
10. There is a history of alcohol abuse, or during the study period the subjects were unable to avoid drinking in the 24 hours before and during the trial drug administration, or those who tested positive for alcohol breath test;
11. There is a history of drug abuse, and the drug screen test results are positive;
12. Blood pregnancy test positive or breastfeeding women;
13. Contraceptives in which the subject or his or her spouse has a family plan within the next 6 months after the last dose and is unable to use research-approved contraceptives during the study period as directed by the investigator;
14. Blood donation or blood loss ≥400 mL in the 3 months before screening, blood donation ≥200 mL in the 1 month before screening;
15. It is impossible to avoid the use of caffeinated beverages, vigorous exercise, or other factors affecting the absorption, distribution, metabolism, and excretion of the drug within 24 hours before and during the trial;
16. Past or existing sick sinus syndrome or other supratrioventricular conduction heart disease such as sinus or atrioventricular block heart disease; Past or existing digestive tract ulcer, bladder outlet obstruction, history of asthma or obstructive pulmonary disease;
17. Participants who have participated or are participating in other clinical trials within 3 months prior to screening;
18. Subjects with other factors deemed unsuitable for participation in this study by the investigator.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 42 days
  AEs and their incidence
Number of Participants With Abnormal Laboratory Values | Up to 42 days
  Number of Participants With Abnormal Laboratory Values
Number of Participants With Abnormal ECG QT Interval | Up to 42 days
  Number of Participants With Abnormal ECG QT Interval
Number of Participants With Abnormal Vital signs | Up to 42 days
  Number of Participants With Abnormal Vital signs
Number of Participants With Abnormal Physical examination | Up to 42 days
  It's comprehensive system check by the doctor.
VAS | Up to 42 days
  Score of Visual Analogue Scale, which is a scale from 0-10, with higher scores indicate more severe.

SECONDARY OUTCOMES:
Cmax of Donepezil | Blood samples collected over a 42-day period
  Maximum observed concentration of drug substance in plasma.
Tmax of Donepezil | Blood samples collected over a 42-day period
  Time when the maximum concentration is acheived
AUC0-t of Donepezil | Blood samples collected over a 42-day period
  Area under the blood concentration-time curve from zero to the collection time t of the last measurable concentration.
AUC0-∞ of Donepezil | Blood samples collected over a 42-day period
  Area under the concentration-time curve from time zero to infinity.
t1/2z of Donepezil | Blood samples collected over a 42-day period
  The time when the concentraion of the drug eliminated to half of the initial.
Vz/F | Blood samples collected over a 42-day period
  Apparent volume of distribution
CLz/F | Blood samples collected over a 42-day period
  Apparent clearance

CONTACTS AND LOCATIONS:
Overall Officials: Dongqing Lv, Principal Investigator — Zhejiang Taizhou Hospital Luqiao Hospital (Enze Hospital)
Locations (1):
- Zhejiang Province Taizhou Hospital Luqiao Hospital (Enze Hospital) (Taizhou Hospital Phase I Center), Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No